CLINICAL TRIAL: NCT05736159
Title: Scientific Justification of Assessment Criteria and Improvement of the Methodology for Assessing School Maturity
Status: Active, not recruiting | Type: Observational
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 020223
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: School Adaptation; School Readiness
Keywords: school maturity; children's health; preventive medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- 3 years old age group: Children from 2 years 10 months 16 days to 3 years 2 months 29 days
  Interventions: Diagnostic Test: Method of assessment of school maturity
- 3.6 years old age group: Children from 3 years 3 months to 3 years 8 months 29 days
  Interventions: Diagnostic Test: Method of assessment of school maturity
- 4 years old age group: Children from 3 years 9 months to 4 years 2 months 29 days
  Interventions: Diagnostic Test: Method of assessment of school maturity
- 4.6 years old age group: Children from 4 years 3 months to 4 years 8 months 29 days
  Interventions: Diagnostic Test: Method of assessment of school maturity
- 5 years old age group: Children from 4 years 9 months to 5 years 2 months 29 days
  Interventions: Diagnostic Test: Method of assessment of school maturity
- 5.6 years old age group: Children from 5 years 3 months to 5 years 8 months 29 days
  Interventions: Diagnostic Test: Method of assessment of school maturity
- 6 years old age group: Children from 5 years 9 months to 6 years 2 months 29 days
  Interventions: Diagnostic Test: Method of assessment of school maturity
- 6.6 years old age group: Children from 6 years 3 months to 6 years 8 months 29 days
  Interventions: Diagnostic Test: Assessment of school adaptation
- 7 years old age group: Children from 6 years 9 months to 7 years 5 months 29 days
  Interventions: Diagnostic Test: Assessment of school adaptation
- 8 years old age group: Children from 7 years 6 months to 8 years 5 months 29 days
  Interventions: Diagnostic Test: Assessment of school adaptation

INTERVENTIONS:
Diagnostic Test: Method of assessment of school maturity — Psychophysiological examination of the functional readiness of the child for admission to school.
  Groups: 3 years old age group; 3.6 years old age group; 4 years old age group; 4.6 years old age group; 5 years old age group; 5.6 years old age group; 6 years old age group
Diagnostic Test: Assessment of school adaptation — Psychophysiological examination of the success of school education of first graders.
  Groups: 6.6 years old age group; 7 years old age group; 8 years old age group

SUMMARY:
One of the critical stages in a child's life is the beginning of school, accompanied by intense intellectual and psycho-emotional stress. The success of educational activities depends on the child's readiness to enter school - his school maturity.

The two main components of school maturity are the level of formation of school skills and the physical development of the child in the preschool period. Recent studies show that adaptation is more favorable in children with an average level of physical development (Zhdanova L.A., Rusova T.V., Shishova A.V., 2020), at the same time there is also a reverse effect - children with a delayed type of development are more susceptible to the development of maladaptation. This relationship opens up new opportunities in the development of methods for assessing school maturity, as well as preventive measures for the timely prevention of maladaptation of children to school.

The relevance of the topic of the peer-reviewed research work is determined by the need to develop and substantiate modern criteria for assessing school maturity.

The purpose of the work is to study the hygienic aspects of children's adaptation to the beginning of school education in order to improve the methodology of comprehensive assessment of school maturity and the development of measures to prevent maladaptation.

To solve it, five tasks have been formulated, the essence of which is to study the factors affecting the course of adaptation of the child, to scientifically substantiate the criteria for assessing school maturity and the development of preventive measures for the timely prevention of maladaptation.

To solve the tasks set, a study of anthropometric indicators and indicators characterizing school maturity and the level of formation of school skills will be conducted among 1,000 children aged 3-8 years studying in preschool educational and general education organizations of the Samara region. The results of the study will be implemented in the work of preschool educational and general education organizations of the Samara region, and in the future, in the department of hygiene of children and adolescents of the Federal Budgetary Health Institution "Center for Hygiene and Epidemiology in the Samara region".

DETAILED DESCRIPTION:
One of the most difficult stages in a child's life is the beginning of school education. Moving from a preschool educational institution to the first grade of school, children face not only intense intellectual loads, but also a change in the daily routine, the need for a long stay at the desk, constant contact with new people, such as classmates and a class teacher.

Under the influence of educational loads, the regulatory system of the body is strained, only a small number of first-graders remain within the limits of the norm - more than a quarter of children are in a state of compensated distress (Ryabova I.V., Filippova S.N., Alekseeva S.I., Sobolevskaya T.A., Chernogorov D.N., 2020).

On how successfully it will pass the period of adaptation of the child depends not only on academic performance, but also on the state of his health and further physical development.

The preschool period has a significant influence on the course of school adaptation. The development of a child at this stage is a predictor of how successful his adaptation to school will be. It is at this age that there is a qualitative change in cognitive functions - memory, voluntary attention, visual perception, as well as the improvement of all types of thinking: logical, visually effective and visually imaginative (Bezrukikh M.M., Filippova T.A., Verba A.S., Ivanov V.V., Sergeeva V.E., 2020). The peculiarities of a child's development at the age of 3-7 years later determine the cognitive, emotional and behavioral components of school adaptation. (Kazakova E.V., Sokolova L.V., 2018).

Therefore, it is necessary to start preparing for school in advance - with an assessment of school maturity and the level of formation of school skills, since the discrepancy between the physical and psychological capabilities of a first-grader to the requirements of the learning environment can lead to the development of maladaptation, negatively affecting all areas and the quality of a child's life.

Determination of children's readiness for school is carried out according to the method of determining the approximate school maturity of Kern-Yirasek, approved in the methodological recommendations of the USSR in 1986. It includes an assessment of the general level of thinking development, the ability to listen and perform tasks according to the sample, as well as hand motor skills and visual perception.

An important role in the adaptation of a child is played by his physical development. Modern research shows that the adaptation process is more favorable for first-graders with an average level of physical development, at the same time there is a feedback: the strain of adaptation contributes to a further slowdown in the pace of child development (Zhdanova L.A., Rusova T.V., Shishova A.V., 2020).

The criterion of the course of adaptation can be distinguished by the dynamics of body weight - during the first quarter of the school year, getting used to new conditions, first-graders are most susceptible to weight loss, and the unfavorable course of adaptation is accompanied by a higher loss of it (Gritsina O.V., Trankovskaya L.V., 2018).

Thus, the relationship between the child's physical development and the course of adaptation opens up new opportunities in the development of methods for assessing the child's school maturity, as well as in the early prevention of maladaptation of schoolchildren. However, this topic requires further in-depth study.

The relevance of the study is connected with the need for scientific substantiation of the criteria for assessing school maturity and the development of preventive measures for the timely prevention of maladaptation of children to school.

The purpose of the study. to study the hygienic aspects of children's adaptation to the beginning of school to improve the methodology of comprehensive assessment of school maturity and the development of measures to prevent maladaptation.

Research objectives.

1. The study of anthropometric indicators and the development of regional age-sex standards of physical development of preschool children.
2. Hygienic assessment of physical development and the level of school maturity of children of older groups of preschool educational organizations and their dynamics during the first grade of school.
3. Identification and scientific substantiation of the factors influencing the process of adaptation of children to schooling.
4. Scientific substantiation of criteria for the development of a methodology for assessing school maturity in preschool children.
5. Development of preventive measures for the timely prevention of maladaptation of children to school.

The candidate's dissertation will be performed as part of a comprehensive research work of the Department of Food Hygiene with the course of hygiene of children and adolescents of the FSBEI HE SamSMU MOH Russia "Hygienic assessment of the impact of factors of conditions and lifestyle on the health of the population of the Samara region".

Object and methods of research. In order to solve the research tasks and obtain reliable results, it is planned to summarize the available data from medical examinations, measure anthropometric indicators and indicators characterizing school maturity and the level of formation of school skills among a representative group of 3-8-year-old children studying in preschool educational and general education organizations of the Samara region. The data obtained will be evaluated using the methods of variational statistics with the determination of the average value, the standard deviation, the error of the average and the determination of the reliability of differences by Student.

Scientific novelty of the research. A comprehensive hygienic assessment of the school adaptation of children and adolescents aged 3-8 years of the Samara region will be carried out at the modern level.

Priority indicators of physical development and school maturity that require management to prevent the development of maladaptation in children of the first grade of education will be determined.

Based on the study of anthropometric indicators, the main regularities of the course of adaptation in first-graders will be established, taking into account their physical development.

Based on the materials received, criteria for assessing the adaptation of first-graders and standards for the physical development of children 3-8 years old in Samara will be developed, as well as hygienic recommendations for preventing the development of maladaptation among children in general education institutions will be substantiated.

Expected results. As a result of the study, indicators will be determined that reliably characterize the level of adaptation of children to school activities.

As a result of the study, indicators will be determined on the basis of which it will be possible to assess the course of adaptation of first-graders of general education organizations of the Samara region.

The results obtained will allow us to develop criteria for assessing the adaptation of first-graders and standards for the physical development of children 3-8 years old, as well as to substantiate hygienic recommendations for preventing the development of maladaptation among children in general education institutions of Samara.

Practical significance of the study. The expected results of the study, as well as the developed hygienic recommendations, can be used by the management of educational institutions, as well as specialists of the Federal Service for Supervision in the Field of Consumer Rights Protection and Human Well-being, who carry out social and hygienic monitoring of environmental factors of children and adolescents.

The level and scope of implementation of the results. The results of the study will be implemented in the work of preschool educational and general education organizations of the Samara region, and in the future, in the department of hygiene of children and adolescents of the Federal Budgetary Health Institution "Center for Hygiene and Epidemiology in the Samara region".

The research materials will be used in conducting practical classes of the discipline "Hygiene of children and adolescents" at the Department of Food Hygiene with the course of hygiene of children and adolescents of the Federal State Budgetary Educational Institution of the Ministry of Health of Russia and in other higher educational medical institutions of Russia.

ELIGIBILITY:
Inclusion Criteria:

* children aged from 3 to 8 years
* first and second health group

Exclusion Criteria:

* diseases in the acute phase

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: Preschool and school-age children
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
the level of adaptation to school | 1/03/2024
  an indicator of the child's adaptation to the conditions of school life, to its norms and requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Regina V. Hamtsova, Principal Investigator — Samara State Medical University
Locations (1):
- SamaraSMU, Samara, Russia